CLINICAL TRIAL: NCT04515108
Title: Comparison of Hematological Parameters and Perinatal Outcomes in COVID-19 Pregnancies and Healthy Pregnancy Cohort
Brief Title: Perinatal Outcomes and Hematologic Parameters in COVID-19 Pregnancies
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Esin Merve Erol Koç, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: E1-20-672
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Pregnancy, Infections in; Covid19
Keywords: COVID-19; Pregnancy; Complete blood count; Perinatal outcome; Monocyte/lymphocyte ratio (MLR)
MeSH Terms: conditions — Pregnancy Complications, Infectious; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Pregnants with COVID-19): Study group included pregnant women with clinically confirmed COVID-19.
  Interventions: Other: Clinical assessment
- Group 2 (Pregnants without COVID-19): Control group consisted of healthy pregnant women in the same number and same gestational week with the Study group.
  Interventions: Other: Clinical assessment

INTERVENTIONS:
Other: Clinical assessment — Perinatal outcomes and diagnostic value of hematologic parameters were compared between pregnancies with and without COVID-19.

SUMMARY:
Complete blood count parameters are routinely evaluated cost-effective markers in diagnosis and clinical follow-up of infectious diseases.There is increasing number of studies to report the course of COVID-19 in pregnancy. The current study aimed to elucidate the changes in hematologic parameters in response to SARS-CoV-2 infection and whether there was an increase in adverse perinatal outcomes such as increased neonatal intensive care unit admission and lower APGAR scores in pregnancies with COVID-19.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the relationship between Coronavirus Disease 2019 (COVID-19) in pregnancy and adverse perinatal outcomes. The secondary aim is to analyze the diagnostic value of hematologic parameters in COVID-19 complicated pregnancies.The current study is conducted in a high volume tertiary obstetrics center burdened by COVID-19 pandemics, in Turkey, between March 20 and July 25, 2020. The study included a pregnant women cohort who had been regularly followed up and delivered in our clinics. The cohort was divided into two groups to reveal the impact of COVID-19 on the complete blood count cell indices and unfavorable obstetric and early neonatal outcomes in pregnant women. The clinically confirmed diagnosis of COVID-19 cases were included in Study Group (n=39) the healthy pregnant women without COVID-19 were included in Control Group (n=69). The study achieved a power of 0.89 and 0.98 with a 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous pregnancy,
* Singleton pregnancy,
* Clinically diagnosed COVID-19 (SARS-CoV-2 positivity in real time-polymerase chain reaction)

Exclusion Criteria:

* Chronic maternal diseases (rheumatological diseases, renal failure, vascular malformations, hypertension, cardiac disease, diabetes mellitus, obesity, hypo-hyperthyroidism, congenital hematological disorders),
* Acute inflammatory conditions (acute pancreatitis, acute appendicitis),
* Pregnancy complications (gestational diabetes, PPROM, preeclampsia),
* Multiple pregnancies,
* Anticoagulant medication.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The current study included 39 pregnant women with clinical diagnosis of COVID-19 on the obstetric isolation unite and 69 pregnant women without COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
complete blood count parameters (including the number of lymphocytes, Leukocytes, monocytes, platelets and red blood cells). | first 1 hour of hospitalization.
  cell count per mm3.

SECONDARY OUTCOMES:
APGAR score | 5 minutes
  1st and 5th minute newborn assessment
maternal and newborn length | 5 minutes
  centimeters
maternal and newborn weight | 2 minutes
  kilograms
body temperature | 2 minutes
  Celsius degree

CONTACTS AND LOCATIONS:
Overall Officials: Esin Merve Erol Koç, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data belonging to participant only will be available to any researcher or editorial review board if needed

REFERENCES:
- [Result] Cheng B, Jiang T, Zhang L, Hu R, Tian J, Jiang Y, Huang B, Li J, Wei M, Yang J, Ren S, Wang G. Clinical Characteristics of Pregnant Women With Coronavirus Disease 2019 in Wuhan, China. Open Forum Infect Dis. 2020 Jul 11;7(8):ofaa294. doi: 10.1093/ofid/ofaa294. eCollection 2020 Aug. PMID 32760752
- [Result] Peng J, Qi D, Yuan G, Deng X, Mei Y, Feng L, Wang D. Diagnostic value of peripheral hematologic markers for coronavirus disease 2019 (COVID-19): A multicenter, cross-sectional study. J Clin Lab Anal. 2020 Oct;34(10):e23475. doi: 10.1002/jcla.23475. Epub 2020 Jul 17. PMID 32681559
- [Result] Sun S, Cai X, Wang H, He G, Lin Y, Lu B, Chen C, Pan Y, Hu X. Abnormalities of peripheral blood system in patients with COVID-19 in Wenzhou, China. Clin Chim Acta. 2020 Aug;507:174-180. doi: 10.1016/j.cca.2020.04.024. Epub 2020 Apr 24. PMID 32339487
- [Result] Dashraath P, Wong JLJ, Lim MXK, Lim LM, Li S, Biswas A, Choolani M, Mattar C, Su LL. Coronavirus disease 2019 (COVID-19) pandemic and pregnancy. Am J Obstet Gynecol. 2020 Jun;222(6):521-531. doi: 10.1016/j.ajog.2020.03.021. Epub 2020 Mar 23. PMID 32217113